CLINICAL TRIAL: NCT05313334
Title: Gamified Approach to Maximizing Biobehavioral Inhibition in Trauma-related Conditions (GAMBIT)
Brief Title: GAMBIT Task With PTSD and Healthy Control Participants
Acronym: GAMBIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study funding not available
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jonathan M DePierro, Associate Professor, Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-01108
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTSD Group (Experimental): The PTSD Group will receive the GAMBIT intervention and complete all study tasks and assessments at every study visit (Visits 0-4). N=20 participants will be recruited for this arm.
  Interventions: Behavioral: GAMBIT Task
- Healthy Control Group (Experimental): The Healthy Control Group will receive the GAMBIT intervention and complete all study tasks and assessments at every study visit (Visits 0-4). N=20 participants will be recruited for this arm. Additionally, N=10 Healthy Control participants will be recruited for the Pilot Phase of the study.
  Interventions: Behavioral: GAMBIT Task

INTERVENTIONS:
Behavioral: GAMBIT Task — The GAMBIT task is a novel inhibitory control task. Participants in the Healthy Control group will receive the GAMBIT intervention repeatedly over the study period.

SUMMARY:
This is a pilot study of a digital training task called GAMBIT. This study will be the first to examine potential relationships between GAMBIT task completion and brain circuit flexibility, behavior, and symptoms in participants with PTSD.

DETAILED DESCRIPTION:
This is a single-site pilot study for the GAMBIT intervention, which is a computerized task that addresses behavioral inhibition. The primary objective of this study is to determine whether the GAMBIT task improves mental health symptoms associated with PTSD over time. The secondary objective of this study is to determine whether the GAMBIT task promotes flexibility in inhibitory control network as determined by functional neuroimaging. Additional laboratory measures associated with cognitive flexibility, and clinician and patient-rated symptom data, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-55 years
* Participants must be able to provide informed consent
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process
* Must meet criteria for one of the following study groups:

  * PTSD Group:

    i. Meets diagnostic criteria for current PTSD according to the Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-5)
    1. Has been exposed to a Criterion A trauma of the civilian type (e.g., non-combat, threatened or actual interpersonal violence) or non-civilian
    2. Must have a total score ≥ 25 on the CAPS-5 (past-month version) at the time of screening, indicating moderate PTSD symptom severity.
  * Healthy Control Group:

    i. Has no lifetime history of any psychiatric disorder

Exclusion Criteria:

* Current or lifetime history of schizophrenia or other psychotic disorder, bipolar disorder, obsessive-compulsive disorder (OCD), eating or feeding disorder, neurodevelopmental disorder, or neurocognitive disorder;
* Any neuropsychiatric disorder that is judged to be the primary presenting problem, other than that which is specified as study group eligibility criteria;
* Substance use disorder within the past 1 year;
* Urine toxicology positive for illicit drugs or dis-allowed concomitant medications as per study protocol; intermittent cannabis use that does not meet criteria for a substance use disorder may be permitted under the protocol.
* Suicidal ideation or risk of self-harm that is judged by the PI to be clinically significant and to warrant intervention
* Concurrent treatment with opioid medication, or with long-acting or daytime short-acting benzodiazepines within two weeks of study start
* Current cognitive impairment, as defined by a score <23 on the Montreal Cognitive Assessment (MoCA)
* Estimated IQ <80
* Currently receiving evidence-based psychotherapy for PTSD (e.g., prolonged exposure, cognitive processing therapy).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) at Baseline | Baseline
  The CAPS is a structured clinical interview designed to assess the essential features of PTSD. A total symptom severity score is calculated on a scale of 0-80, with a higher score representing greater symptom severity.
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) at Day 23 | Day 23
  The CAPS is a structured clinical interview designed to assess the essential features of PTSD. A total symptom severity score is calculated on a scale of 0-80, with a higher score representing greater symptom severity.
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) at Day 52 | Day 52
  The CAPS is a structured clinical interview designed to assess the essential features of PTSD. A total symptom severity score is calculated on a scale of 0-80, with a higher score representing greater symptom severity.

SECONDARY OUTCOMES:
Inhibitory Control Network Flexibility at Baseline | Baseline
  Network flexibility will be determined from resting state FMRI-derived metrics using relatively novel statistical techniques.
Inhibitory Control Network Flexibility at Day 52 | Day 52
  Network flexibility will be determined from resting state FMRI-derived metrics using relatively novel statistical techniques.
PTSD Checklist for DSM-5 (PCL-5) at Baseline | Baseline
  The PTSD Checklist for DSM-5 (PCL-5) is a widely used clinical self-report scale to evaluate current symptoms of PTSD. Each question on the 20-item checklist corresponds to a symptom of PTSD in the DSM-5. A total severity score is calculated on a scale of 0-80, with a higher score indicating greater severity.
PTSD Checklist for DSM-5 (PCL-5) Weekly for Weeks 1-6 | Weekly [Weeks 1-6]
  The PTSD Checklist for DSM-5 (PCL-5) is a widely used clinical self-report scale to evaluate current symptoms of PTSD. Each question on the 20-item checklist corresponds to a symptom of PTSD in the DSM-5. A total severity score is calculated on a scale of 0-80, with a higher score indicating greater severity.
PTSD Checklist for DSM-5 (PCL-5) at Day 23 | Day 23
  The PTSD Checklist for DSM-5 (PCL-5) is a widely used clinical self-report scale to evaluate current symptoms of PTSD. Each question on the 20-item checklist corresponds to a symptom of PTSD in the DSM-5. A total severity score is calculated on a scale of 0-80, with a higher score indicating greater severity.
PTSD Checklist for DSM-5 (PCL-5) at Day 52 | Day 52
  The PTSD Checklist for DSM-5 (PCL-5) is a widely used clinical self-report scale to evaluate current symptoms of PTSD. Each question on the 20-item checklist corresponds to a symptom of PTSD in the DSM-5. A total severity score is calculated on a scale of 0-80, with a higher score indicating greater severity.
Combined Think/No-Think and Go/No-Go Paradigm | up to 52 days
  The combined Think/No-Think and Go/No-Go paradigm requires participants to learn 35 cue-target word pairs (for approximately 15 minutes) and then asked to alternatively suppress, recall, or think about the cue-target word pairs, when prompted. The percentage of correctly processed trials (go/think trials and no-go/no-think trials) are calculated per block, on a scale from 0% (0/35 trials) to 100% (35/35 trails), with higher recall scores on no-go/no-think trials indicating worse inhibitory control.
Face-Stroop Task | up to 52 days
  The Face-Stroop task is a modified version of the widely used Stroop task which assesses reaction time between congruent and incongruent stimuli. During the Face-Stroop task, participants are simultaneously presented with images of emotional faces and emotional words (e.g., "Happy", "Sad"), with some trials presenting congruent stimuli (happy face + "Happy") and other trials presenting incongruent stimuli (happy face + "Sad"), and asked to identify the faces and words separately. Variables of interest include reaction time (range 250-1000 milliseconds, with lower RT indicating better performance) and accuracy (0-100%, with greater accuracy denoting better performance).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan DePierro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.

DOCUMENTS (1):
  • Informed Consent Form (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT05313334/ICF_000.pdf